CLINICAL TRIAL: NCT04615325
Title: A Phase 1a, Multicenter, Open-label, Single-dose, Dose-escalation Study of the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Intravitreal Injections of RO7303359 in Patients With Geographic Atrophy Secondary to Age-related Macular Degeneration
Brief Title: A Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Intravitreal Injections of RO7303359 in Participants With Geographic Atrophy Secondary to Age-related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GR42163
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Single Ascending Dose Stage (Experimental): Participants will receive a single dose of RO7303359, in multiple escalating cohorts (A-D).
  Interventions: Drug: RO7303359
- Expansion Cohort Stage (Experimental): Participants will receive the maximum tolerated dose (MTD) or the maximum tested dose (MTeD) as determined in the single ascending dose stage.
  Interventions: Drug: RO7303359
- Optional Cohort E (Experimental): An optional additional cohort may be added with the dose not exceed the MTD or MTeD.
  Interventions: Drug: RO7303359
- Optional cohort F (Experimental): An optional additional cohort may be added with the dose not exceed the MTD or MTeD.
  Interventions: Drug: RO7303359

INTERVENTIONS:
Drug: RO7303359 — RO730359 will be administered as a single intravitreal injection.

SUMMARY:
This multicenter study will investigate the safety, tolerability, pharmacokinetics, and immunogenicity of RO7303359 following single intravitreal (ITV) injection in participants with geographic atrophy (GA) secondary to age-related macular degeneration (AMD). Participants will receive an ITV injection of RO7303359 in the single ascending dose stage and the maximum tolerated dose (MTD) or maximum tested dose (MTeD) of RO7303359 in the expansion stage.

ELIGIBILITY:
Ocular Inclusion Criteria Study Eye:

* Visual acuity: BCVA letter score of 19-48 ETDRS letters (Snellen equivalent of 20/125-20/400) using ETDRS charts at a starting distance of 4 meters
* Well-demarcated area of GA secondary to AMD in the absence of choroidal neovascularization (CNV)
* GA area must be >/= 0.5 disc area (1.25 mm^2)

Ocular Exclusion Criteria, Study Eye:

* GA in the study eye due to causes other than AMD
* History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD
* Previous laser photocoagulation for CNV, diabetic macular edema, retinal vein occlusion, or proliferative diabetic retinopathy
* Prior treatment with photodynamic therapy, external beam radiation therapy (for intraocular conditions), or transpupillary thermotherapy

Ocular Exclusion Criteria, Both eyes:

* Evidence of prior or active CNV
* Previous participation in interventional clinical trials for GA or dry AMD, except for vitamins and minerals, irrespective of the route of administration (i.e. ocular or systemic) within the last 6 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Ocular Adverse Events | Up to 12 weeks
Percentage of Participants With Systemic Adverse Events | Up to 12 weeks
Percentage of Participants With Dose-limiting Adverse Events (DLAEs), | Up to 12 weeks
Percentage of Participants With Serious Adverse Events (SAEs) | Up to 12 weeks
Percentage of Participants With Adverse Events Leading to Study Discontinuation | Up to 12 weeks
Percentage of Participants With Adverse Events of Special Interest (AESIs) | Up to 12 weeks
Change from Baseline in Best Corrected Visual Acuity (BCVA) Score as Assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) Chart | Baseline, Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- United States (12):
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retinal Consultants Med Group, Sacramento, California
  - California Retina Consultants - Santa Maria, Santa Maria, California
  - Colorado Retina Associates, PC, Denver, Colorado
  - Florida Eye Associates, Melbourne, Florida
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Associated Retinal Consultants PC, Royal Oak, Michigan
  - Sierra Eye Associates, Reno, Nevada
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Tennessee Retina PC., Nashville, Tennessee
  - Austin Clinical Research LLC, Austin, Texas
  - Retina Foundation of the Southwest, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Pearlman JA, Sheth VS, Khanani AM, Indjeian VB, Brunstein F, Kuruvilla D, Maia M, Dere R, Ma L, Chen H, Datta S, Willis JR, Wiley HE. Phase I Study of the Anti-interleukin 33 Fragment Antigen-Binding Region RO7303359 in Geographic Atrophy Secondary to Age-Related Macular Degeneration. Ophthalmol Sci. 2025 Apr 20;5(5):100800. doi: 10.1016/j.xops.2025.100800. eCollection 2025 Sep-Oct. PMID 40538770